CLINICAL TRIAL: NCT02374684
Title: A Within-group Randomized, Double-Blind, Placebo-Controlled, Single/ Multiple Dose Study to Assess the Safety , Tolerability, Pharmacokinetics and Food Effect of Methosulide After Oral Administration In Healthy Adult Subjects.
Brief Title: Tolerability, Safety and Pharmacokinetic Study Of Methosulide in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hubei Biological Medicine Industrial Technology Institute Co., Ltd. (Other)
Collaborators: Academy Military Medical Science, China (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HubeiBMITI- CM2010-01-I
Record Dates: First submitted 2015-02-05; First posted 2015-03-02 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
Keywords: Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methosulide (Experimental): Methosulide, oral administration
  Interventions: Drug: Methosulide
- Placebo (Placebo Comparator): Placebo, oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methosulide — Tolerability Study:
  Period I:Single oral administration,dose-escalation of Methosulide(six dose groups:25mg-250mg) Period II:Repeated oral administration of Methosulide(group 1:MTD（maximum tolerated dose）/250mg ,group 2:depending on the adverse drug reaction,150mg/250mg)
  Pharmacokinetic Study:
  Period I:Single oral administration,dose-escalation of Methosulide(three dose groups:50mg,100mg,200mg/250mg) Period II:Repeated oral administration of Methosulide(group 1:MTD（maximum tolerated dose）/250mg
  ,group 2:depending on the adverse drug reaction,150mg/250mg)
  Food Effect on the Pharmacokinetics:
  single dose(100mg),two status(Feeding and fasting), washout period(7 days)
  Other Names: CM2010-01
  Arms: Methosulide
Drug: Placebo — Placebo to match with experimental groups
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and tolerability, and to evaluate the pharmacokinetic characteristics and food effect of Methosulide after oral administration in healthy adult subjects.

DETAILED DESCRIPTION:
1. Dose-escalation study of single oral administration of Methosulide in healthy adults to assess the safety and tolerability.
2. Multiple-dose study of Methosulide in healthy adults to assess the safety and tolerability.
3. Dose-escalation study of single oral administration of Methosulide in healthy adults to evaluate the pharmacokinetic characteristics
4. Multiple-dose study of Methosulide in healthy adults to evaluate the pharmacokinetics characteristics
5. Single dose,and cross-over study of Methosulide in healthy adults to evaluate the pharmacokinetic characteristics and effect of food.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between 18 and 45 years of age, Body Mass Index (BMI) between 19～25 kg/m2, Weight > or = 50kg
* In good health as judged by the investigator
* Without history of medication within 2 weeks before the test
* Non-allergic constitution, without known drug allergy
* Without history of major organ diseases
* Without other factors affecting drug metabolism, such as smoking (within 2 weeks), drinking (within 2 weeks), or drug abuse history
* Signed informed consent form and Fully understood the contents, process and possible adverse reactions of the test

Exclusion Criteria:

* History of kinds of food or drug allergy, or suffering from allergic diseases or allergic constitution
* Presence (in screening stage) or history of the acute/chronic organic diseases or clinical manifestations: blood system, renal disease, endocrine system, respiratory system, digestive system, cardiovascular system, nervous system, mental disease, allergic diseases (including drug allergy, but not including non-treatment, asymptomatic, seasonal allergy during the period of oral administration)
* History of abuse of Smoking, alcohol, or other drugs
* Severe hemorrhage factors to affect the venous blood collection
* Severe blood loss or blood donation within 3 months before the test
* Participation in other drug trials within 3 months before the test
* Usage of drugs known to have damage to the main organs within 3 months before the test
* Without good compliance, or unable to match with the test
* with a clinically significant abnormality in routine serological detection: including Hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) infected
* For childbearing-aged women only, usage of any hormonal contraceptive methods within 3 months before the drug administration; or unable or unwilling to use non-hormonal contraceptive methods to contraception from the day of dosing until 14 days after dosing
* Be otherwise unsuitable for the study, in the opinion of the Investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2015-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single and repeated oral administration of Methosulide as measured by the frequency of drug-related clinical adverse events in healthy adults. | Period I: single dose,Baseline - 7 Days;Period II: repeated dose,Baseline - 14 Days
  Adverse events, vital signs, electrocardiograms, physical exams, and clinical laboratory assessments will be assessed prior to, during, and after treatment

SECONDARY OUTCOMES:
Cmax of single oral administration of Methosulide and effect of food in healthy adults. | Baseline - 7 Days
Tmax of single oral administration of Methosulide and effect of food in healthy adults. | Baseline - 7 Days
area under curve(AUC) of single oral administration of Methosulide and effect of food in healthy adults. | Baseline - 7 Days
t1/2α of single oral administration of Methosulide and effect of food in healthy adults. | Baseline - 7 Days
t1/2β of single oral administration of Methosulide and effect of food in healthy adults. | Baseline - 7 Days
Vd of single oral administration of Methosulide and effect of food in healthy adults. | Baseline - 7 Days
Cls of single oral administration of Methosulide and effect of food in healthy adults. | Baseline - 7 Days
Css of repeated oral administration of Methosulide in healthy adults. | Baseline - 14 Days
Cmax of repeated oral administration of Methosulide in healthy adults. | Baseline - 14 Days
Tmax of repeated oral administration of Methosulide in healthy adults. | Baseline - 14 Days
area under curve(AUC) of repeated oral administration of Methosulide in healthy adults. | Baseline - 14 Days
t1/2α of repeated oral administration of Methosulide in healthy adults. | Baseline - 14 Days
t1/2β of repeated oral administration of Methosulide in healthy adults. | Baseline - 14 Days
Vd of repeated oral administration of Methosulide in healthy adults. | Baseline - 14 Days
Cls of repeated oral administration of Methosulide in healthy adults. | Baseline - 14 Days

CONTACTS AND LOCATIONS:
Overall Officials: ZHENG Heng, Principal Investigator — Tongji Hospital, Affiliated to Tongji Medical College of Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan，Hubei, China